CLINICAL TRIAL: NCT04611451
Title: Effect of Whole Body Vibration Exercises for Patients wıth Chronic Nonspeific Low Back Pain on Labor and Quality of Life: a Randomized Controlled Trial
Brief Title: Effect of Whole Body Vibration Exercises for Patients wıth Chronic Nonspeific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yerkoy State Hospital (Other)
Responsible Party: Principal Investigator, Başak Çiğdem Karaçay, specialist, Yerkoy State Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/70
Record Dates: First submitted 2020-10-20; First posted 2020-11-02 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Pain; Labor Pain; Quality of Life; Disability Physical
Keywords: low back pain; whole body vibration; labor
MeSH Terms: conditions — Pain; Labor Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration group (Experimental): Patients in the WBV exercise group; 24 sessions of TVT exercise 3 days a week (with at least 1 day of rest between each session) was performed under the supervision of a physician for a total of 8 weeks. Patients in the WBV exercise group were also shown a classic lumbar home exercise program and they were asked to apply for 8 weeks
  Interventions: Other: classic lumbar home exercise; Device: Whole body vibration; Other: Whole body vibration exercise
- exercise (Active Comparator): The second group (control) only received classical lumbar home exercise program.
  Interventions: Other: classic lumbar home exercise

INTERVENTIONS:
Other: classic lumbar home exercise — classic lumbar home exercise
Device: Whole body vibration — Whole body vibration (WBV), which is a new treatment method and applied through the device, is defined as mechanical repetitive motion or oscillatory motion occurring around a balance point
  Arms: whole body vibration group
Other: Whole body vibration exercise — Whole body vibration exercise
  Arms: whole body vibration group

SUMMARY:
Whole body vibration (WBV), which is a new treatment method and applied through the device, is defined as mechanical repetitive motion or oscillatory motion occurring around a balance point (5). Chronic nonspecific low back pain is still a serious clinical, social and economic health problem. There are few studies and limited evidence evaluating the effectiveness of WBV exercises in chronic nonspecific low back pain. Different protocols are used for wbv exercise in studies (6). Our aim is to compare the effects of whole body vibration exercise modality on pain, functional recovery, laboor impact, quality of life with control group in patients with chronic nonspecific low back pain.

DETAILED DESCRIPTION:
Low back pain is a prevalent problem all over the World. low back pain prevalence is 84% by lifetime Chronic low back pain prevalence is 23%. Low back pain causing disability prevalence is also11% (1). Increasing sedentary lifestyle and obesity, aging of the population and inappropriate ergonomic work activities and working environment in the working society contribute to this increase (2).

Chronic low back pain is an important cause of labor losses and also it is the most common functional insufficiency under 45 years of age (3). Treatment approaches such as exercise and education in which the patient is actively involved in the treatment are recommended for the treatment of non-specific acute, subacute and especially chronic low back pain (4).

Whole body vibration (WBV), which is a new treatment method and applied through the device, is defined as mechanical repetitive motion or oscillatory motion occurring around a balance point (5). Chronic nonspecific low back pain is still a serious clinical, social and economic health problem. There are few studies and limited evidence evaluating the effectiveness of WBV exercises in chronic nonspecific low back pain. Different protocols are used for wbv exercise in studies (6). Our aim is to compare the effects of whole body vibration exercise modality on pain, functional recovery, laboor impact, quality of life with control group in patients with chronic nonspecific low back pain.

MATERYAL METHOD

This prospective, randomized and controlled study include 70 patients who were diagnosed chronic nonspecific low back pain. Patients were randomized into two groups using the 1:1 method. The first group was the treatment group in which applied the whole body vibration exercise and classical lumbar home exercise program. The second group (control) only received classical lumbar home exercise program.

Inclusion criterias are non-specific LBP (LBP other than those excluded, see exclusion criteria below) of a more than 3 months in patients aged 20 to 50 years, with average pain intensity evaluated Visaual Analog Scale (VAS) (1-10) that is higher than 5 Exclusion criterias are participants with likely specific causes of LBP This includes exclusion of history of malignancy, history of recent spinal surgery, dislocation, fracture, rheumatoid arthritis and ankylosing spondylitis and history of weakness of lower extremity or loss of sensation in lower extremity. Additionally, current pregnancy, , lactation, uncontrolled hypertension and history of diagnosed mental health conditions that would limit adherence to the trial procedures will be excluded.

Patients in the TVT exercise group; 24 sessions of TVT exercise 3 days a week (with at least 1 day of rest between each session) was performed under the supervision of a physician for a total of 8 weeks. . The vibration was given by the Power Plate® (pro5TM; Power Plate North America, Inc., Northbrook, IL, USA) device where a three-plan oscillation took place (most vertical, Z-axis).The Istanbul Low Back Pain Disability index is a self-reported measure of functional disability . The Istanbul Low Back Pain Disability index has reliability and validit(7). Quality of life was assessed using Short form-36 (SF-36). SF-36 is a widely used and validated scale in assessing quality of life. It is not specific to any disease group. Health and Labor Questionnaire (HLQ) was used in our study to evaluate job performance. HLQ is designed to collect quantitative data on the treatment of disease and its relationship to work performance. Intercultural adaptation was made to Turkish. HLQ data allow to estimate the production losses (costs) of paid and unpaid labor (8).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criterias are non-specific LBP (LBP other than those excluded, see exclusion criteria below) of a more than 3 months in patients aged 20 to 50 years, with average pain intensity evaluated Visaual Analog Scale (VAS) (1-10) that is higher than 5

Exclusion Criteria:

* Exclusion criterias are participants with likely specific causes of LBP This includes exclusion of history of malignancy, history of recent spinal surgery, dislocation, fracture, rheumatoid arthritis and ankylosing spondylitis and history of weakness of lower extremity or loss of sensation in lower extremity. Additionally, current pregnancy, , lactation, uncontrolled hypertension and history of diagnosed mental health conditions that would limit adherence to the trial procedures will be excluded

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 20-50 years old
Enrollment: 70 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Health and Labor Questionnaire (HLQ) | baseline (0 day)
  Health and Labor Questionnaire (HLQ) was used in our study to evaluate job performance. HLQ is designed to collect quantitative data on the treatment of disease and its relationship to work performance. Intercultural adaptation was made to Turkish. HLQ data allow to estimate the production losses (costs) of paid and unpaid labor
Health and Labor Questionnaire (HLQ) | 8 week
  Health and Labor Questionnaire (HLQ) was used in our study to evaluate job performance. HLQ is designed to collect quantitative data on the treatment of disease and its relationship to work performance. Intercultural adaptation was made to Turkish. HLQ data allow to estimate the production losses (costs) of paid and unpaid labor
Health and Labor Questionnaire (HLQ) | 20 week
  Health and Labor Questionnaire (HLQ) was used in our study to evaluate job performance. HLQ is designed to collect quantitative data on the treatment of disease and its relationship to work performance. Intercultural adaptation was made to Turkish. HLQ data allow to estimate the production losses (costs) of paid and unpaid labor
Quality of life Short form-36 (SF-36) | baseline (0 day)
  Quality of life was assessed using Short form-36 (SF-36). SF-36 is a widely used and validated scale in assessing quality of life. It is not specific to any disease group. This scale consisting of 36 questions; It has 8 subgroups as general health, physical function, physical role difficulty, pain, energy, social function, emotional role difficulty, mental health.
Quality of life Short form-36 (SF-36) | 8 week
  Quality of life was assessed using Short form-36 (SF-36). SF-36 is a widely used and validated scale in assessing quality of life. It is not specific to any disease group. This scale consisting of 36 questions; It has 8 subgroups as general health, physical function, physical role difficulty, pain, energy, social function, emotional role difficulty, mental health.
Quality of life Short form-36 (SF-36) | 20 week
  Quality of life was assessed using Short form-36 (SF-36). SF-36 is a widely used and validated scale in assessing quality of life. It is not specific to any disease group. This scale consisting of 36 questions; It has 8 subgroups as general health, physical function, physical role difficulty, pain, energy, social function, emotional role difficulty, mental health.
Visual Analog Scale | baseline (0 day)
  Visual Analog Scale was used for pain
Visual Analog Scale | 8 week
  Visual Analog Scale was used for pain
Visual Analog Scale | 20 week
  Visual Analog Scale was used for pain

SECONDARY OUTCOMES:
disability | baseline (0 day)
  The Istanbul Low Back Pain Disability index is a self-reported measure of functional disability consisting of 18 questions about various activities related to back pain. Each question has 6 possible responses ranging from 0 to 5, with a total possible maximum score of 50. The total Istanbul Low Back Pain Disability index score is with higher percentages indicating greater levels of self-reported disability. The Istanbul Low Back Pain Disability index has reliability and validit(7).
disability | 8 week
  The Istanbul Low Back Pain Disability index is a self-reported measure of functional disability consisting of 18 questions about various activities related to back pain. Each question has 6 possible responses ranging from 0 to 5, with a total possible maximum score of 50. The total Istanbul Low Back Pain Disability index score is with higher percentages indicating greater levels of self-reported disability. The Istanbul Low Back Pain Disability index has reliability and validit(7).
disability | 20 week
  The Istanbul Low Back Pain Disability index is a self-reported measure of functional disability consisting of 18 questions about various activities related to back pain. Each question has 6 possible responses ranging from 0 to 5, with a total possible maximum score of 50. The total Istanbul Low Back Pain Disability index score is with higher percentages indicating greater levels of self-reported disability. The Istanbul Low Back Pain Disability index has reliability and validit(7).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Weiner SS, Nordin M. Prevention and management of chronic back pain. Best Pract Res Clin Rheumatol. 2010 Apr;24(2):267-79. doi: 10.1016/j.berh.2009.12.001. PMID 20227647
- [Background] Ladeira CE. Evidence based practice guidelines for management of low back pain: physical therapy implications. Rev Bras Fisioter. 2011 May-Jun;15(3):190-9. doi: 10.1590/s1413-35552011000300004. PMID 21829982
- [Background] Sitja Rabert M, Rigau Comas D, Fort Vanmeerhaeghe A, Santoyo Medina C, Roque i Figuls M, Romero-Rodriguez D, Bonfill Cosp X. Whole-body vibration training for patients with neurodegenerative disease. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD009097. doi: 10.1002/14651858.CD009097.pub2. PMID 22336858
- [Background] Perraton L, Machotka Z, Kumar S. Whole-body vibration to treat low back pain: fact or fad? Physiother Can. 2011 Winter;63(1):88-93. doi: 10.3138/ptc.2009.44. Epub 2011 Jan 20. PMID 22210985
- [Background] Duruoz MT, Ozcan E, Ketenci A, Karan A. Development and validation of a functional disability index for chronic low back pain. J Back Musculoskelet Rehabil. 2013;26(1):45-54. doi: 10.3233/BMR-2012-00349. PMID 23411648
- [Background] McGorry RW, Webster BS, Snook SH, Hsiang SM. The relation between pain intensity, disability, and the episodic nature of chronic and recurrent low back pain. Spine (Phila Pa 1976). 2000 Apr 1;25(7):834-41. doi: 10.1097/00007632-200004010-00012. PMID 10751295
- [Background] cakar E, Özcan E, Özgörgü E, Durmuş O, Karan A, Kıralp MZ. Health and labour questionnaire: Turkish adaptation for ankylosing spondylitis. Türk Fiz Tıp Rehab Derg. 2012;58(3):205-12.